CLINICAL TRIAL: NCT03234608
Title: Health System Integration of Tools to Improve Primary Care for Autistic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland State University (Other)
Collaborators: Oregon Health and Science University (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Christina Nicolaidis, Professor, Portland State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34MH111536-01 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-31 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Healthcare services; Adults
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: We will conduct the study in primary care clinics within three health systems. We will compare data from patients in 7 intervention clinics to patients from matched control clinics within the same systems.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AASPIRE Healthcare Toolkit (Experimental): Patients will use the AASPIRE Healthcare Toolkit and will share a copy of their Autism Healthcare Accommodations Report with their primary care provider.
  Interventions: Behavioral: AASPIRE Healthcare Toolkit
- Usual Care (No Intervention): Patients will receive usual care.

INTERVENTIONS:
Behavioral: AASPIRE Healthcare Toolkit — The AASPIRE Healthcare Toolkit includes a variety of resources (information, worksheets, checklists, links) for patients and providers. The centerpiece of the toolkit is the Autism Healthcare Accommodations Tool, which allows a patient or their supporter to create a personalized accommodations report for the patient's provider. Intervention patients will use the toolkit and create an AHAT report. Intervention clinics will receive a copy of each patient's AHAT report, place it in the medical record, and share it with the patient's PCP and other staff.
  Arms: AASPIRE Healthcare Toolkit

SUMMARY:
The health system is ill-equipped to meet the needs of autistic adults. The Academic Autism Spectrum Partnership in Research and Education (AASPIRE), an academic-community partnership comprised of academics, autistic adults, healthcare providers, and supporters, has used a community based participatory research (CBPR) approach to develop and test an online healthcare toolkit aimed at improving primary care services for autistic adults. It was specifically designed as a low-intensity, sustainable intervention that can realistically be used in busy primary care practices that do not have a special focus on autism or other developmental disabilities. The toolkit includes the Autism Healthcare Accommodations Tool (AHAT)--an automated tool which allows patients and/or their supporters to create a personalized accommodations report for their primary care provider (PCP)--and other targeted resources, worksheets, checklists, and information. The investigators' pilot work has demonstrated that the AHAT has strong construct validity and test-retest stability, the toolkit is highly acceptable and accessible, and it has the potential to decrease barriers to care and increase patient-provider communication. The investigators' long-term plan is to conduct a hybrid effectiveness-implementation trial, using a cluster randomized trial design, both to test the effectiveness of the AASPIRE Healthcare Toolkit in improving healthcare quality and utilization and to assess the utility of implementation strategies in diverse healthcare systems. The objective of this proposal is to use a CBPR approach to understand how to integrate the toolkit into these health systems, collect more robust efficacy data, and explore potential mechanisms of action. The investigators will do so by conducting a 6-month pilot study with patients assigned to intervention and control clinics in three diverse health systems. The investigators will meet our objectives by achieving the following specific aims: 1) to determine how to integrate use of the toolkit within diverse health systems; 2) to test the effect of the toolkit on short-term healthcare outcomes; 3) to use a mixed-methods approach to further explore the toolkit's mechanisms of action; and 4) to refine the recruitment, retention, data collection, and system integration strategies in preparation for the larger cluster-randomized trial.

DETAILED DESCRIPTION:
Despite growing attention to the needs of autistic children, the health system is ill equipped to meet the needs of autistic adults. The investigators' prior work has identified significant healthcare disparities experienced by autistic adults, including greater unmet healthcare needs, lower use of preventive services, and greater use of the Emergency Department (ED). These disparities likely stem from a complex interaction between patient-, provider-, and system-level factors. Autism entails atypical communication and interpersonal relationships, and challenges with executive function - factors that are critically important for effective healthcare interactions and health system navigation. Moreover, a majority of primary care providers (PCPs) lack the skills needed to care for autistic adults, yet competing priorities make it unlikely they will attend trainings on autism. The heterogeneity of the autism spectrum may also make it challenging to understand a specific patient's needs. Finally, autistic patients may be disproportionally affected by the complexity of the health system, low socio-economic status, and societal biases, yet few systems can afford autism-specific care coordination programs for adults.

The Academic Autism Spectrum Partnership in Research and Education (AASPIRE), an academic-community partnership comprised of academics, autistic adults, healthcare providers, and supporters, has used a community based participatory research (CBPR) approach to develop and test an online healthcare toolkit aimed at improving primary care services for autistic adults. It was specifically designed as a low-intensity, sustainable intervention that can realistically be used in busy primary care practices that do not have a special focus on autism or other developmental disabilities. The toolkit includes the Autism Healthcare Accommodations Tool (AHAT)--an automated tool which allows patients and/or their supporters to create a personalized accommodations report for their PCP--and other targeted resources, worksheets, checklists, and information. A series of NIMH-funded studies demonstrated that the AHAT has strong construct validity and test-retest stability, and that the toolkit is highly acceptable and accessible. In a 1-month pre-post intervention comparison, the investigators found a decrease in barriers to care and increases in patient-provider communication and confidence in healthcare. Despite these promising preliminary results, more data is needed to test its effectiveness and understand how to best integrate it into diverse primary care practices and health systems.

The investigators' long-term plan is to conduct a hybrid effectiveness-implementation trial, using a cluster randomized trial design, both to test the effectiveness of the AASPIRE Healthcare Toolkit in improving healthcare quality and utilization and to determine the potential utility of implementation strategies in diverse healthcare systems. The objective of this proposal is to use a CBPR approach to understand how to best integrate the toolkit into these health systems, collect more robust efficacy data, and explore potential mechanisms of action. The investigators will do so by conducting a 6-month pilot study with patients assigned to intervention and control clinics in three diverse health systems. The investigators will meet our objectives by achieving the following specific aims:

1. To determine how to integrate use of the toolkit within diverse health systems. The investigators' existing CBPR partnership will expand to include local patients, providers, staff, and administrators from each system. Together, the investigators will decide how to make patients and providers aware of the toolkit, integrate the AHAT into the electronic medical record, and respond to recommendations. The investigators will collaboratively develop implementation protocols and determine how to track them. The investigators will then conduct a mixed-methods, formative process evaluation to optimize the likelihood of success of future implementation efforts.'
2. To test the effect of the toolkit on short-term healthcare outcomes. The investigators hypothesize that, over 6 months, the toolkit will increase satisfaction with patient-provider communication and decrease barriers to healthcare in patients from intervention clinics as compared to patients from control clinics.
3. To use a mixed-methods approach to further explore the toolkit's mechanisms of action. Quantitative data will help the investigators refine and psychometrically test our measures of patient self-advocacy and visit preparedness; provider/staff use of desired accommodations and strategies; and patient and provider self-efficacy. Qualitative data will allow the investigators to obtain a richer understanding of how the toolkit is affecting care and potentially suggest additional mechanisms of action.
4. To refine our recruitment, retention, data collection, and system integration strategies in preparation for the larger cluster-randomized trial. The investigators will use this study to confirm or modify our change model, choose long-term health utilization outcomes to be further studied in the R01, finalize study protocols and data collection instruments, and develop a flexible implementation strategy that can be feasibly applied to diverse primary care clinics.

Successful integration of this scalable and sustainable low-intensity intervention into primary care practices within diverse health systems will empower patients and providers to work together to improve health outcomes for a large, underserved and understudied population with great barriers to care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic code in chart related to autism spectrum disorder or other communication disability
* Receiving care at one of participating clinics

Exclusion Criteria:

* Can neither participate directly (with or without support), nor has an English-speaking supporter who can answer surveys on their behalf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Nicolaidis, MD, MPH, Principal Investigator — Portland State University
Locations (3):
- United States (3):
  - Kaiser Permanente Northern California, Oakland, California
  - Legacy Health System, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Participating in National Institute of Mental Health (NIMH) Data Archive
Supporting Information: Study Protocol
Time Frame: After study completion.
Access Criteria: Determined by NIMH Data Archive

RESULTS

PARTICIPANT FLOW:
Groups:
- AASPIRE Healthcare Toolkit: Patients will use the Academic Autism Spectrum Partnership in Research and Education (AASPIRE) Healthcare Toolkit and will share a copy of their Autism Healthcare Accommodations Tool (AHAT) Report with their primary care provider.
  AASPIRE Healthcare Toolkit: The AASPIRE Healthcare Toolkit includes a variety of resources (information, worksheets, checklists, links) for patients and providers. The centerpiece of the toolkit is the Autism Healthcare Accommodations Tool, which allows a patient or their supporter to create a personalized accommodations report for the patient's provider. Intervention patients will use the toolkit and create an AHAT report. Intervention clinics will receive a copy of each patient's AHAT report, place it in the medical record, and share it with the patient's Primary Care Provider (PCP) and other staff.
Period: Overall Study
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
Started | 127 | 117
Completed | 104 | 96
Not Completed | 23 | 21
Not completed — Lost to Follow-up | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care | Total
Number analyzed (Participants) | 127 | 117 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.32 (12.86) | 29.03 (10.94) | 30.22 (12.01)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Participants with complete data
  Participants
    Gender: number analyzed (Participants) | 125 | 116 | 241
    Gender: Male | 82 | 86 | 168
    Gender: Female | 39 | 29 | 68
    Gender: Other | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants with complete data
  Participants
    number analyzed (Participants) | 124 | 115 | 239
    Non-Hispanic White | 80 | 67 | 147
    Non-Hispanic Black / African-American | 7 | 17 | 24
    Non-Hispanic Asian / Pacific Islander | 8 | 10 | 18
    Non-Hispanic Multi-Racial | 14 | 8 | 22
    Hispanic or Latino | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  United States | 127 | 117 | 244
Participant Residence [Count of Participants; unit: Participants] — Population: Participants with complete data
  Participants
    number analyzed (Participants) | 124 | 115 | 239
    Place they own or rent | 47 | 27 | 74
    With family | 74 | 87 | 161
    Group home/Foster home | 0 | 0 | 0
    Other | 3 | 1 | 4
Participant need assistance from someone for medical care [Count of Participants; unit: Participants] — Population: Participants with complete data
  Participants
    number analyzed (Participants) | 114 | 107 | 221
    Always or often | 45 | 41 | 86
    Sometimes | 31 | 21 | 52
    Rarely or never | 38 | 45 | 83
Participant help with communication [Count of Participants; unit: Participants] — Population: Participants with complete data
  Participants
    number analyzed (Participants) | 123 | 115 | 238
    Communicate with providers by themselves | 57 | 47 | 104
    Someone helps them some of the time | 45 | 33 | 78
    Someone does most or all of the communication | 21 | 35 | 56
Participant overall health [Count of Participants; unit: Participants] — Population: Participants with complete data
  Participants
    number analyzed (Participants) | 124 | 115 | 239
    Poor | 6 | 4 | 10
    Fair | 19 | 19 | 38
    Good | 40 | 38 | 78
    Very good | 37 | 41 | 78
    Excellent | 22 | 13 | 35
Patient-Provider Communication Scale (PPCS-8) [Mean (Standard Deviation); unit: units on a scale] — AASPIRE Patient-Provider Communication Scale (PPCS-8): This scale is scored by summing responses to the 8 items. Scores range from 8 to 40, with higher scores indicating higher satisfaction with patient-provider communication. Population: Participants with complete data
  units on a scale
    number analyzed (Participants) | 124 | 111 | 235
    (all) | 32.76 (5.71) | 33.14 (5.83) | 32.94 (5.76)
The AASPIRE Visit Preparedness Scale (VPS-6) [Mean (Standard Deviation); unit: units on a scale] — AASPIRE Visit Preparedness Scale (VPS-6): The scale is scored by summing responses to the 6 items. It has a range of 6-30, with higher scores indicating higher visit preparedness. This scale measures how well-prepared patient felt for their most recent visit. Population: Participants with complete data
  units on a scale
    number analyzed (Participants) | 121 | 112 | 233
    (all) | 23.80 (3.76) | 23.90 (4.13) | 23.85 (3.93)
Barriers to Healthcare Checklist-Short Form [Mean (Standard Deviation); unit: units on a scale] — Barriers to Healthcare Checklist-Short Form: The instrument is scored as a count of the total number of barriers endorsed from a checklist of 16 items. Scores can range from 0 to 16. The score depicts the number of barriers to healthcare the participants reports. Higher scores depict a worse outcome. Population: Participants with complete data
  units on a scale
    number analyzed (Participants) | 123 | 116 | 239
    (all) | 2.63 (3.08) | 2.19 (2.34) | 2.42 (2.75)
Healthcare Accommodations Scale(HAS-8) [Mean (Standard Deviation); unit: units on a scale] — AASPIRE Healthcare Accommodations Scale (HAS-8): The scale is scored by summing responses from the eight items. The resulting scale can range from 8 to 40, with higher scores indicating higher receipt of necessary accommodations. Patient report, using 8-item scale, of how well clinic providers and staff make necessary accommodations. Population: Participants with complete data
  units on a scale
    number analyzed (Participants) | 118 | 107 | 225
    (all) | 28.88 (6.00) | 29.84 (6.27) | 29.34 (6.14)
Individual Level Healthcare Self Efficacy Sub-scale [Mean (Standard Deviation); unit: units on a scale] — AASPIRE Health and Healthcare Self-Efficacy Scale (HHSES-21): This is a 21-item scale about patient confidence in navigating the healthcare system and managing health problems. There are two sub-scales. The Individual Level Self-Efficacy Sub-scale consists of items 1, 2, 3, 4, 11, 13,14, 15, 16, and 17. It is scored by summing responses to the items, and then dividing the sum by the number of items (10). The resulting sub-scale has a possible range of 1-10, with higher scores corresponding to higher self-efficacy. Population: Participants with complete data
  units on a scale
    number analyzed (Participants) | 126 | 113 | 239
    (all) | 7.51 (1.67) | 7.72 (1.52) | 7.61 (1.60)
Relationship-Dependent Healthcare Self-Efficacy Sub-scale [Mean (Standard Deviation); unit: units on a scale] — AASPIRE Health and Healthcare Self-Efficacy Scale (HHSES-21): This is a 21-item scale about patient confidence in navigating the healthcare system and managing health problems. There are two sub-scales. The Relationship Dependent Self-Efficacy Sub-scale consists of items 5, 6, 7, 8, 9, 10, 12, 18, 19, 20, and 21. It is scored by summing responses to the items, and then dividing the sum by the number of items (11). The resulting sub-scale has a possible range of 1-10, with higher scores corresponding to higher self-efficacy. Population: Participants with complete data
  units on a scale
    number analyzed (Participants) | 126 | 113 | 239
    (all) | 7.26 (1.89) | 7.49 (1.82) | 7.37 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in Barriers to Healthcare
Description: Barriers to Healthcare Checklist-Short Form: The instrument is scored as a count of the total number of barriers endorsed from a checklist of 16 items. Scores can range from 0 to 16. The score depicts the number of barriers to healthcare the participants reports. A higher number of barriers is a worse outcome.
  Change in barriers to healthcare is calculated by subtracting the baseline score from the 6 month score. Negative scores depict an improvement (i.e. participant is reporting fewer barriers 6 months after the intervention than they did at baseline).
Time Frame: Baseline and 6 months
Population: Participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
Number analyzed (Participants) | 102 | 91
units on a scale | -0.44 (1.92) | -0.42 (2.07)
Statistical Analysis 1: Comparison: AASPIRE Healthcare Toolkit vs Usual Care; Test type: Superiority; p = 0.56, Regression, Linear — The threshold for statistical significance was p<0.05; Slope = 0.18, 95% CI 2-sided [-0.44 to 0.81], Standard Error of Mean 0.32

2. Primary Outcome: Change in Patient-Provider Communication
Description: AASPIRE Patient-Provider Communication Scale (PPCS-8): This scale is scored by summing responses the 8 items. Scores range from 8 to 40, with higher scores indicating higher satisfaction with patient-provider communication.
  Change in patient-provider communication is calculated by subtracting the score at baseline from the score at 6 months. Positive scores indicate an improved outcome (i.e. better patient-provider communication post-intervention than before).
Time Frame: Baseline and 6 months
Population: Participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
Number analyzed (Participants) | 99 | 89
units on a scale | -0.49 (5.26) | -0.48 (4.86)
Statistical Analysis 1: Comparison: AASPIRE Healthcare Toolkit vs Usual Care; Test type: Superiority; p = 0.73, Regression, Linear — The threshold for statistical significance was p<0.05; Slope = 0.28, 95% CI 2-sided [-1.28 to 1.84], Standard Error of Mean 0.79

3. Secondary Outcome: Change in Healthcare Self-Efficacy
Description: AASPIRE Health and Healthcare Self-Efficacy Scale (HHSES-21): This is a 21-item scale about patient confidence in navigating the healthcare system and managing health problems. There are two sub-scales. The Individual Level Self-Efficacy Sub-scale consists of items 1, 2, 3, 4, 11, 13,14, 15, 16, and 17. The Relationship Dependent Self-Efficacy Sub-scale consists of items 5, 6, 7, 8, 9, 10, 12, 18, 19, 20, and 21. Each sub-scale is scored by summing responses to the items, and then dividing the sum by the number of items. The resulting sub-scales have a possible range of 1-10, with higher scores corresponding to higher self-efficacy.
  Change in healthcare self-efficacy is calculated by subtracting the baseline score from the score at 6 months. A positive score indicates an improved outcome (i.e. higher self-efficacy post-intervention).
Time Frame: Baseline and 6 months
Population: Participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
Number analyzed (Participants) | 103 | 92
units on a scale
  Individual Level Self-Efficacy Sub-scale | 0.11 (1.10) | 0.06 (1.06)
  Relationship Dependent Self-Efficacy Sub-scale | 0.19 (1.30) | 0.08 (1.45)
Statistical Analysis 1: Comparison: AASPIRE Healthcare Toolkit vs Usual Care; Statistical analysis for Individual Level Healthcare Self-Efficacy Sub-scale; Test type: Superiority; p = 0.94, Regression, Linear — The threshold for statistical significance was p<0.05; Slope = -0.01, 95% CI 2-sided [-0.35 to 0.33], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: AASPIRE Healthcare Toolkit vs Usual Care; Statistical analysis for Relationship-Dependent Healthcare Self-Efficacy Sub-scale; Test type: Superiority; p = 0.65, Regression, Linear; Slope = 0.10, 95% CI 2-sided [-0.33 to 0.52], Standard Error of Mean 0.21

4. Secondary Outcome: Change in Visit Preparedness
Description: AASPIRE Visit Preparedness Scale (VPS-6): The scale is scored by summing responses to the 6 items. It has a range of 6-30, with higher scores indicating higher visit preparedness. This scale measures how well-prepared patient felt for their most recent visit.
  Change in visit preparedness is calculated by subtracting the baseline score from the score at 6 months. Positive scores indicate an improved outcome (i.e. higher visit preparedness post-intervention).
Time Frame: Baseline and 6 months
Population: Participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
Number analyzed (Participants) | 98 | 91
units on a scale | -0.04 (3.17) | 0.05 (3.21)
Statistical Analysis 1: Comparison: AASPIRE Healthcare Toolkit vs Usual Care; Test type: Superiority; p = 0.66, Regression, Linear — The threshold for statistical significance was p<0.05; Slope = -0.23, 95% CI 2-sided [-1.25 to 0.79], Standard Error of Mean 0.52

5. Secondary Outcome: Change in Receipt of Healthcare Accommodations
Description: AASPIRE Healthcare Accommodations Scale (HAS-8): The scale is scored by summing responses from the eight items. The resulting scale can range from 8 to 40, with higher scores indicating higher receipt of necessary accommodations. Patient report, using 8-item scale, of how well clinic providers and staff make necessary accommodations.
  Change in receipt of healthcare accommodations is calculated by subtracting the baseline score from the score at 6 months. A positive change in score indicates an improved outcome (i.e. greater receipt of necessary accommodations after the intervention).
Time Frame: Baseline and 6 months
Population: Participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
Number analyzed (Participants) | 94 | 87
units on a scale | 0.80 (5.10) | -0.07 (4.38)
Statistical Analysis 1: Comparison: AASPIRE Healthcare Toolkit vs Usual Care; Test type: Superiority; p = 0.85, Regression, Linear — The threshold for statistical significance was p<0.05; Slope = 0.15, 95% CI 2-sided [-1.40 to 1.69], Standard Error of Mean 0.78

6. Other Pre Specified Outcome: Healthcare Use
Description: Patient self-report of use of preventive, outpatient, and emergency services; unmet healthcare needs
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Satisfaction With Healthcare Toolkit
Description: Open- and closed-ended survey and interview questions about patient satisfaction with healthcare toolkit (intervention only)
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Provider Confidence and Satisfaction
Description: Survey items on primary care provider's confidence in caring for autistic patients and satisfaction with toolkit
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events reported during the duration of the study.
Arm/Group | AASPIRE Healthcare Toolkit | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/117
Other Adverse Events (participants affected / at risk) | 0/127 | 0/117

LIMITATIONS AND CAVEATS:
This study aimed to integrate the AASPIRE Healthcare Toolkit into 3 healthcare systems. The intervention relied on primary care providers receiving and using a patients' Autism Healthcare Accommodations Report (AHAT). Unfortunately, due to various implementation challenges, very few providers received the AHAT reports. As such, most participants in the intervention arm did not receive the intended intervention. Data cannot be used to assess intervention efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03234608/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03234608/ICF_001.pdf